CLINICAL TRIAL: NCT05629936
Title: Improving Medication Therapy and Patient Involvement Through a Digital Interdisciplinary Model Among Old People in Primary Care Living in Sparsely Populated Regions in Sweden
Brief Title: Improving Medication Therapy Through a Digital Interdisciplinary Medicine Therapy Optimisation Model
Acronym: MTO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Maria Gustafsson, Principal investigator, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UMU-MTO-2022
Record Dates: First submitted 2022-11-07; First posted 2022-11-29 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Drug Use
Keywords: Telemedicine; Medication reconciliation; Clinical pharmacist; Elderly; Adherence; Drug-related problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital intervention (Other): Digital intervention
  Interventions: Other: Digital interdisciplinary intervention

INTERVENTIONS:
Other: Digital interdisciplinary intervention — Digital medication interview, comprehensive medication review, interdisciplinary patient-centred discussions, follow-ups

SUMMARY:
This study investigates if a digital interdisciplinary medicine therapy optimisation (MTO) model in primary care can improve medication therapy, quality of life, medication adherence, and beliefs about medicines, among patients >65 years living in sparsely populated areas. The intervention includes digital medication interviews, comprehensive medication reviews, interdisciplinary patient-centred discussions, and follow-ups.

DETAILED DESCRIPTION:
Initially, a pilot study will be conducted to evaluate the feasibility of the method and to make appropriate adjustments to the study design before starting the main study. Patients that meet the inclusion criteria will be invited to participate in the study via letter. The patients will also receive three validated questionnaires; Medication Adherence Report Scale-5 (MARS-5), EuroQol-5 Dimension-5 Level questionnaire (EQ-5D-5L) and The Beliefs about Medicines Questionnaire (BMQ) to fill in prior to initiation of the study, to collect baseline data. The intervention consists of several steps and all meetings are digital. At first, the patient will have a medication interview with a clinical pharmacist, Next, the clinical pharmacist conducts a comprehensive medication review based on information from the interview and the participant's medical records and laboratory values. The clinical pharmacist and the participant's primary care physician will then have a joint discussion regarding preliminary medication management proposals and therapy management plans. The patient will be informed by their physician if any medication changes have been made. Digital follow-up meetings with the patient and the clinical pharmacist will take place 1-2, 4 and 12 weeks after the baseline consultation, and additionally if requested by the patient or if the pharmacist consider it necessary. The clinical pharmacist will also conduct repeated medical record reviews every second week during the 12-week intervention period. After the last follow-up at 12 weeks, the patient will be asked to fill in the three questionnaires: MARS-5, EQ-5D-5L and BMQ one more time.

ELIGIBILITY:
Inclusion Criteria:

* Using 5 or more medications or recommended by the primary care physician (e.g. according to the use of certain medicines or conditions such as chronic kidney disease)
* Living at home (i.e not in a nursing home)
* Registered at certain primary healthcare centres in the rural areas of Västerbotten

Exclusion Criteria:

* Do not speak Swedish or unable to communicate
* Has home care services
* Has a confirmed major neurocognitive disorder
* Receives palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification and resolution of drug-related problems | The 12-week intervention period
  Categorisation of drug-related problems according to a modified version of the Cipolle-Strand-Morley criteria 2012
Change in self-reported medication adherence: Medication Adherence Report Scale-5 (MARS-5) | Baseline and 12 weeks
  Assessing self-reported medication adherence through the MARS-5 questionnaire. Total score ranging between 5 and 25, with higher scores indicating a higher level of medication adherence.
Change in self-reported health-related quality of life: EuroQol-5 Dimension-5 Level questionnaire (EQ-5D-5L) | Baseline and 12 weeks
  Assessing health-related quality of life through the EQ-5D-5L-questionnaire. The questionnaire consists of five questions regarding self-perceived quality of life, and a visual analogue scale on which the respondents evaluate their own health status on a scale of 0-100.
Change in self-reported beliefs about medicines: The Beliefs about Medicines Questionnaire (BMQ) | Baseline and 12 weeks
  Assessing beliefs about medicines through BMQ. The questionnaire consists of two different scales; BMQ-General assesses the respondent's beliefs about drugs in general and BMQ-Specific evaluates the individual's beliefs about medicines prescribed for their own use.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gustafsson, Ph.D, Principal Investigator — Department of Medical and Translational Biology, Umeå University
Locations (1):
- Storuman healthcare centre, Storuman, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Westberg A, Andersson P, Sonnerstam E, Mattsson S, Holmner A, Edin-Liljegren A, Gustafsson M. Development and evaluation of a telepharmacy service in primary care for home-living older adults in Northern Sweden's rural areas: protocol for a single-arm interventional study. BMJ Open. 2025 Nov 19;15(11):e110198. doi: 10.1136/bmjopen-2025-110198. PMID 41263936